CLINICAL TRIAL: NCT04775849
Title: Intraoperative Berger Space Imaging
Brief Title: Intraoperative Berger Space Imaging (IBSI)
Acronym: IBSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Menapace, Clinical Professor, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IBSI - 2258/2018
Record Dates: First submitted 2021-02-23; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Cataract; Macula Edema
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Cataract surgery will be performed in individuals with age-related cataract.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoperative Berger Space Imaging (Experimental): Intraoperative OCT imaging of the space between the posterior capsule and the anterior hyaloid
  Interventions: Device: Femtosecond Laser

INTERVENTIONS:
Device: Femtosecond Laser — Femtosecond Laser assisted Cataract Surgery will be performed uni- or bilateral

SUMMARY:
The investigational device is an approved femtosecond laser (FSL) device with an integrated imaging system to perform certain steps of the cataract procedure. The FSL will perform anterior capsulotomy and lens fragmentation in individuals suffering from age-related cataract with need of cataract surgery.

The laser will be reduced to image the Berger space. If not visible, the space will be enhanced with BSS and Volon A to visualize the BS.

Cataract surgery will be performed in subjects who have signed an informed consent form. Macula thickness will be measured with Spectralis OCT on screening date.

Postoperative examinations will be implemented in accordance with the approved investigational plan on subjects and includes: visual acuity, slitlamp examination and retinal oct imaging.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral age-related cataract necessitating phacoemulsification extraction and posterior IOL implantation
* Age: 40 to 90 (females of childbearing age will be interviewed if pregnancy is possible)
* Preoperative pupil size in mydriasis ≥ 6.0 mm

Exclusion Criteria:

* Preceding ocular surgery or trauma
* Pseudoexfoliation
* Recurrent intraocular inflammation of unknown etiology
* Uncontrolled glaucoma
* Uncontrolled systemic or ocular disease
* Blind fellow eye
* Microphthalmus
* Corneal abnormality
* History of uveitis/iritis
* Iris neovascularization
* Proliferative diabetic retinopathy
* Macular degeneration or any other relevant macular diseases
* Pregnancy

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
The primary objective is a Berger Space larger than 400μm | intraoperative
  The number of patients with visible Berger space and the capacity (volume) of the visible Berger Space will be determined by using the intraoperative OCT recording

SECONDARY OUTCOMES:
Difference of central macular thickness between time points | Baseline to 1day, 1 week, 3 weeks
  Difference in Central Macular Thickness (CMT) with time.
Intraocular pressure in different timepoints | Baseline to 1day, 1 week, 3 weeks
  Intraocular pressure changes with time.

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Menapace, MD, Principal Investigator — Medical Universitiy of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No